CLINICAL TRIAL: NCT04050553
Title: A Randomized, Placebo-Controlled, Crossover Study to Investigate the Effect of Once-Weekly Tirzepatide on the Counter-Regulatory Response to Hypoglycemia in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17222; I8F-MC-GPHG (Other: Eli Lilly and Company); 2019-001360-29 (EudraCT Number)
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Experimental): Participants received a starting dose of 2.5 mg tirzepatide once weekly (QW) for 2 weeks, followed by an increase to 5 mg QW for 2 weeks, and 10 mg QW for 4 weeks until the 15-mg dose was reached and maintained for the remainder of the treatment period (4 weeks) administered subcutaneously (SC) in one of two study periods.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants received placebo QW administered SC in one of two study periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about how tirzepatide affects the body's response to low blood sugar (hypoglycemia). The study is open to participants with type 2 diabetes. It will last about 42 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) for at least 1 year
* Treated with diet and exercise and stable dose(s) of metformin 3 months prior to study entry with or without 1 additional oral antidiabetic medication (OAM) other than metformin.
* Have a hemoglobin A1c (HbA1c) value at screening of ≥6.5% and ≤9.0 % if on metformin only.
* Have a HbA1c value at screening of ≥6.0% and ≤8.5 %, if on metformin and 1 more allowed OAM.
* Have a body mass index (BMI) between 23 and 45 kilograms per square meter (kg/m²) inclusive, at screening
* Are of stable weight (±5%) >3 months prior to screening

Exclusion Criteria:

* Have a history of proliferative retinopathy or maculopathy as determined by the investigator based on a recent (<6 months) ophthalmologic examination
* Impaired renal estimated glomerular filtration rate (eGFR) <60 milliliters per minute per 1.73 square meters (mL/min/1.73 m²) calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data
* Have had acute myocardial infarction, congestive heart failure New York Heart Association Class III or IV, history of or suspected ischemic heart disease, and/or cerebrovascular accident (stroke [including transient ischemic attack])

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Universitätsklinikum Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieber TR, Svehlikova E, Urva S, Haupt A, Zhou C, Coskun T, Holler V, Fluhr G, Karanikas CA, Milicevic Z, Pratt EJ. Counterregulatory response to hypoglycemia during a hypoglycemic clamp in people with type 2 diabetes treated with tirzepatide. Front Endocrinol (Lausanne). 2025 Sep 2;16:1627947. doi: 10.3389/fendo.2025.1627947. eCollection 2025. PMID 40964167

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Tirzepatide 15 Milligrams (mg): Period 1: Participants received placebo administered subcutaneously (SC) once-weekly (QW) for 12 weeks; Wash-out: 8-10 weeks; Period 2: Participants received a starting dose of 2.5 mg tirzepatide given SC QW for 2 weeks, followed by an increase to 5 mg QW for 2 weeks, and 10 mg QW for 4 weeks until the 15-mg dose was reached and maintained for the remainder of the treatment period (4 weeks).
- Tirzepatide 15 mg/Placebo: Period 1: Participants received a starting dose of 2.5 mg tirzepatide given SC QW for 2 weeks, followed by an increase to 5 mg QW for 2 weeks, and 10 mg QW for 4 weeks until the 15-mg dose was reached and maintained for the remainder of the treatment period (4 weeks); Wash-out: 8-10 weeks; Period 2: Participants received placebo administered SC QW for 12 weeks.
Period: Period 1
Arm/Group | Placebo/Tirzepatide 15 Milligrams (mg) | Tirzepatide 15 mg/Placebo
Started | 21 | 21
Received At Least One Dose of Study Drug | 21 | 21
Completed | 18 | 17
Not Completed | 3 | 4
Not completed — Physician Decision | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Wash-out
Arm/Group | Placebo/Tirzepatide 15 Milligrams (mg) | Tirzepatide 15 mg/Placebo
Started | 18 | 17
Completed | 18 | 15
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Placebo/Tirzepatide 15 Milligrams (mg) | Tirzepatide 15 mg/Placebo
Started | 18 | 15
Received At Least One Dose of Study Drug | 18 | 15
Completed | 18 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo/Tirzepatide 15 mg: Period 1: Participants received placebo administered SC QW for 12 weeks; Wash-out: 8-10 weeks; Period 2: Participants received a starting dose of 2.5 mg tirzepatide given SC QW for 2 weeks, followed by an increase to 5 mg QW for 2 weeks, and 10 mg QW for 4 weeks until the 15-mg dose was reached and maintained for the remainder of the treatment period (4 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo/Tirzepatide 15 mg | Tirzepatide 15 mg/Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (4.8) | 55.4 (7.4) | 57.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 19 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Glucagon Concentration During Induced Hypoglycemia From Target Plasma Glucose (PG) Concentration of 100 Milligrams Per Deciliter (mg/dL) to a Nadir Target of 45 mg/dL
Description: A linear mixed effects model, with treatment, treatment period, and treatment sequence as fixed effects, and patient as a random effect using restricted maximum likelihood (REML) method was used. PG of plateau 100 mg/dL was considered as baseline timepoint.
Time Frame: Week 12 in each study period: Baseline and up to 30 minutes after reaching the nadir glucose level.
Population: All participants who received at least one dose of study drug and had evaluable Pharmacodynamic (PD) data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: picomole per liter (pmol/L)
Groups:
- Placebo: Participants received placebo administered SC QW for 12 weeks.
- Tirzepatide 15 mg: Participants received a starting dose of 2.5 mg tirzepatide given SC QW for 2 weeks, followed by an increase to 5 mg QW for 2 weeks, and 10 mg QW for 4 weeks until the 15-mg dose was reached and maintained for the remainder of the treatment period (4 weeks).
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 32 | 33
picomole per liter (pmol/L) | 18.55 (1.64) | 18.07 (1.62)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; Test type: Superiority; p = 0.7556, Mixed Models Analysis; Least Square (LS) Mean Difference = -0.49, 95% CI 2-sided [-3.64 to 2.67]

2. Secondary Outcome: Change in Mean Insulin Concentrations From Induced Hypoglycemia Target PG Concentration of 100 mg/dL to a Nadir Target of 45 mg/dL
Description: A linear mixed effects model, with treatment, treatment period, and treatment sequence as fixed effects, and patient as a random effect using REML method was used.
Time Frame: Week 12 in each study period: Baseline and up to 30 minutes after reaching the nadir glucose level.
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: picomole per liter (pmol/L)
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 32 | 33
picomole per liter (pmol/L) | -1053.31 (54.20) | -1228.08 (53.61)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; Test type: Superiority; p = 0.0043, Mixed Models Analysis; LS Mean Difference = -174.77, 95% CI 2-sided [-290.34 to -59.21]

3. Secondary Outcome: Change in Mean C-peptide Concentrations From Induced Hypoglycemia Target PG Concentration of 100 mg/dL to a Nadir Target of 45 mg/dL
Description: as for outcome 2
Time Frame: Week 12 in each study period: Baseline and up to 30 minutes after reaching the nadir glucose level.
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: picomole per liter (pmol/L)
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 32 | 33
picomole per liter (pmol/L) | -177.69 (51.78) | -665.99 (51.09)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -488.31, 95% CI 2-sided [-621.25 to -355.36]

4. Secondary Outcome: Time From Termination of Insulin Infusion at PG Concentration of 45 mg/dL to Reach Recovery PG Concentration (72 mg/dL)
Description: as for outcome 2
Time Frame: Week 12 in each treatment period (treatment period = 12 weeks): 1 minute after reaching the nadir glucose level and when reaching normoglycemia (estimated as 30 mins).
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: minutes (min)
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 31 | 32
minutes (min) | 43.34 (1.29) | 47.73 (1.27)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; Test type: Superiority; p = 0.0023, Mixed Models Analysis; LS Mean Difference = 4.39, 95% CI 2-sided [1.69 to 7.08]

5. Secondary Outcome: Hypoglycemia Symptoms Score From Induced Hypoglycemia at Target PG Concentrations of 100 mg/dL, 63 mg/dL, 45 mg/dL and Recovery (PG Concentration 72 mg/dL)
Description: Hypoglycemia symptoms score was measured with the Edinburgh Hypoglycemia Symptom Scale (EHSS) which is a 13-item questionnaire for hypoglycemic symptoms: 10 neuroglycopenic symptoms (6 cognitive dysfunctions: inability to concentrate, blurred vision, anxiety, confusion, difficulty speaking, and double vision; 4 neuroglycopenia: drowsiness, tiredness, hunger, and weakness), and 3 autonomic symptoms (sweating, trembling, and warmness) and participants were asked to rate the intensity of their hypoglycemic symptoms on a 7-point Likert scale (1 = No symptom to 7 = Severe). The total score is the sum of scores from the 13 questions and ranged from 13 to 91. This score was scaled back to the range of 1 to 7 by taking average of the sum of scores (i.e., sum of the scores divided by number of questions), where lower score indicates fewer symptoms.
Time Frame: Week 12.
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 33 | 33
Score on a scale
  100 mg/dL | 1.19 (0.03) | 1.13 (0.03)
  63 mg/dL | 1.35 (0.06) | 1.17 (0.06)
  45 mg/dL: number analyzed (Participants) | 31 | 33
  45 mg/dL | 1.68 (0.08) | 1.49 (0.08)
  72 mg/dL | 1.50 (0.09) | 1.38 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; For Overall Hypoglycemia Symptom Score at concentration of 100 mg/dL; Test type: Superiority; p = 0.0505, Mixed Models Analysis; LS Mean Difference = -0.06, 95% CI 2-sided [-0.13 to 0.00]
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide 15 mg; For Overall Hypoglycemia Symptom Score at concentration of 63 mg/dL; Test type: Superiority; p = 0.0104, Mixed Models Analysis; LS Mean Difference = -0.18, 95% CI 2-sided [-0.31 to -0.05]
Statistical Analysis 3: Comparison: Placebo vs Tirzepatide 15 mg; For Overall Hypoglycemia Symptom Score at concentration of 45 mg/dL; Test type: Superiority; p = 0.0068, Mixed Models Analysis; LS Mean Difference = -0.19, 95% CI 2-sided [-0.32 to -0.06]
Statistical Analysis 4: Comparison: Placebo vs Tirzepatide 15 mg; For Overall Hypoglycemia Symptom Score at concentration of 72 mg/dL; Test type: Superiority; p = 0.2302, Mixed Models Analysis; LS Mean Difference = -0.11, 95% CI 2-sided [-0.30 to 0.08]

6. Secondary Outcome: Mean Change in Blood Pressure From Induced Hypoglycemia Target PG Nadir Concentration of 100 mg/dL to a Nadir Target of 45 mg/dL
Description: as for outcome 2
Time Frame: Week 12 in each study period: Baseline and up to 30 minutes after reaching the nadir glucose level.
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury (mmHg)
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 31 | 33
millimeters of Mercury (mmHg)
  Systolic Blood Pressure | -5.01 (2.22) | -5.51 (2.17)
  Diastolic Blood Pressure | -9.84 (1.16) | -7.88 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; For systolic blood pressure; Test type: Superiority; p = 0.8298, Mixed Models Analysis; LS Mean Difference = -0.51, 95% CI 2-sided [-5.28 to 4.27]
Statistical Analysis 2: Comparison: Placebo vs Tirzepatide 15 mg; For diastolic blood pressure; Test type: Superiority; p = 0.1516, Mixed Models Analysis; LS Mean Difference = 1.96, 95% CI 2-sided [-0.76 to 4.67]

7. Secondary Outcome: Mean Change in Heart Rate From Induced Hypoglycemia Target PG Concentration of 100 mg/dL to a Nadir Target of 45 mg/dL
Description: as for outcome 2
Time Frame: Week 12 in each study period: Baseline and up to 30 minutes after reaching the nadir glucose level.
Population: All participants who received at least one dose of study drug and had evaluable PD data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (beats/min)
Arm/Group | Placebo | Tirzepatide 15 mg
Number analyzed (Participants) | 31 | 33
beats per minute (beats/min) | 5.56 (1.26) | 4.67 (1.23)
Statistical Analysis 1: Comparison: Placebo vs Tirzepatide 15 mg; Test type: Superiority; p = 0.5776, Mixed Models Analysis; LS Mean Difference = -0.89, 95% CI 2-sided [-4.10 to 2.33]

ADVERSE EVENTS:
Time Frame: Baseline Through End of Safety Follow-Up (Up To 36 Weeks)
Description: All participants who received at least one dose of study drug. Per protocol, Adverse Event analysis was planned as per treatment regimen received.
Arm/Group | Placebo | Tirzepatide 15 mg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/36 | 4/39
Other Adverse Events (participants affected / at risk) | 13/36 | 27/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Tirzepatide 15 mg (N=39)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | Tirzepatide 15 mg (N=39)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 4 (5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Eructation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 15 (27)
Vomiting (Gastrointestinal disorders) | 1 (2) | 6 (8)
Injection site reaction (General disorders) | 0 (0) | 3 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Pancreatic enzymes increased (Investigations) | 1 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 7 (9)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT04050553/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04050553/SAP_001.pdf